CLINICAL TRIAL: NCT03336385
Title: The Influence of Prebiotic Supplementation on Intestinal Barrier Function in Elderly: A Randomized Placebo Controlled Clinical Trial
Brief Title: Prebiotic Supplementation and Intestinal Barrier Function in Elderly: a RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Örebro University, Sweden (Other)
Collaborators: Fibebiotics consortium (EU) (Unknown)
Responsible Party: Principal Investigator, Robert Brummer, Professor, MD, Örebro University, Sweden
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: FIT
Record Dates: First submitted 2017-09-14; First posted 2017-11-08 (Actual); Last update posted 2018-08-23 (Actual); Status verified 2018-08

CONDITIONS: Prebiotics; Aged
Keywords: Older adults; Prebiotics; Intestinal permeability; NSAIDS

STUDY DESIGN:
Intervention Model Description: The study participants were allocated through block randomization into three different intervention arms that ran in parallell throughout the study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The randomization list was generated and provided by the Fibebiotics consortium (part of the EU framework 7 program) using unique study codes for participants.
  All study product labels were coded by a third-party. All investigators and study participants remained blinded until final analysis
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Maltodextrin 12 gram used as placebo
  Interventions: Dietary Supplement: Placebo
- Naxus (Active Comparator): Naxus contains the wheat-derived prebiotic fibre Arabinoxylan
  Interventions: Dietary Supplement: Naxus
- Oatwell (Active Comparator): Oatwell contains an oat-derived prebiotic beta-glucan fibre
  Interventions: Dietary Supplement: Oatwell

INTERVENTIONS:
Dietary Supplement: Naxus — Non-digestible polysaccharides arabinoxylan (Naxus)
  Other Names: Placebo
  Arms: Naxus
Dietary Supplement: Oatwell — Non-digestible polysaccharides oat beta-glucan (Oatwell)
  Arms: Oatwell
Dietary Supplement: Placebo — Maltodextrin as placebo
  Arms: Placebo

SUMMARY:
The investigators aim was to assess whether 6 weeks of oral intake of the wheat-derived prebiotic fiber arabinoxylan or oat-derived beta-glucan could improve intestinal barrier function against drug-induced barrier disruption in a general population of elderly people, in a randomized double blinded placebo-controlled clinical trial.

DETAILED DESCRIPTION:
The study consisted of a 9 week clinical trial to which the study participants orally ingested two different prebiotic compounds/one placebo for a total of 6 weeks.

The primary outcome was intestinal permeability which was measured before/after indomethacin intake before starting with the prebiotic supplementation and repeated 6 weeks afterwards.

Indomethacin is an NSAID known to artificially increase the intestinal permeability. The prebiotic fibers arabinoxylan and oat-derived beta-glucan have not been investigated for their effect on intestinal permeability in older adults.

Intestinal permeability was investigated using the multi-sugar permeability test. Participants ingested a water solution containing 5 sugar probes that are taken up in different parts of the gut. These sugars are later recovered in the urine at two different time points, reflecting gastroduodenal, small intestinal and colonic permeability.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent signed by study participant
* Age ≥ 55 years
* Mentally and physically fit to complete questionnaires during the study period

Exclusion Criteria:

* Known or genic gastrointestinal disease, with strictures, malignance's and ischemia.
* Inflammatory bowel diseases (IBD)
* Participation in other clinical trials in the past three months.
* Intake of medications know to change the inflammatory status (i.e proton pump inhibitors, antibiotic, anti-inflammatory medication (including NSAIDs)

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-10-12 (Actual); Primary Completion 2015-12-18 (Actual); Study Completion 2015-12-18 (Actual)

PRIMARY OUTCOMES:
Changes in delta indomethacin challenged permeability at end of intervention period | 6 weeks
  In vivo multi-sugar permeability test

SECONDARY OUTCOMES:
Changes in faecal microbiota composition at end of intervention period | 6 weeks
  16S rRNA-based sequencing
Changes in cytokine levels at end of intervention period | 6 weeks
  Multiplex assay for IL-1β, IL-6, IL-8, IL-10, IL-2, IL-12p70, IFN-γ and TNF-α
Changes in reactive oxygen species levels at end of intervention period | 6 weeks
  FORT test for hydrogen peroxide
Changes in gastrointestinal symptom questionnaire scores at end of intervention period | 6 weeks
  The Gastrointestinal Symptoms Rating Scale (GSRS) evaluates gastrointestinal (GI) symptoms based on the 5 domains diarrhoea, constipation, reflux, indigestion and abdominal pain. The symptoms are assessed with 15 items, ranging in scores 1 to 7 depending on their severity. A score of 1 represents "no problems" and score 7 represents "severe problems". The severity of symptoms may be defined as no problems (1 point), mild (1-2 points), moderate (2-4 points), and severe (4-7 points). The scores for each domain was calculated as the mean score of each corresponding item while the mean total GSRS score reflects the general severity of GI symptoms.
Changes in hospital and anxiety depression scores at end of intervention period | 6 weeks
  The Hospital Anxiety and Depression Scale (HADS) was used to evaluate the psychological distress of study participants.This questionnaire consists of 14 items subdivided in two subscales for the assessment of anxiety or depression. The total score is used as a measure of general psychological distress. The minimum score is 0 and the maximum score is 21. A score > 8 on respective subscales indicates a significant level of anxiety or depression.
Changes in perceived stress scale scores at end of intervention period | 6 weeks
  The perceived stress scale (PSS) consists of 10 items, including a number of direct questions about current levels of experienced stress. The respondent answers how often a certain emotion has been present during the past month. PSS scores are obtained by reversing responses (e.g., 0 = 4, 1 = 3, 2 = 2, 3 = 1 & 4 = 0) to the four positively stated items (items 4, 5, 7, & 8) and then summing across all scale items. Each item is rated on a 5-point scale ranging from never (0) to almost always (4). The questions in this scale ask about the responders feelings and thoughts during the last month. In each case the questionnaire requires the respondent to indicate by circling how often they felt or thought a certain way.
Changes in quality of life questionnaire scores at end of intervention period | 6 weeks
  The EuroQol 5D-5L (EQ-5D-5L) tool consists of two parts; 5Q-5D, which includes 5 items related to wellbeing and function (mobility, self-care, usual activities, pain/discomfort and anxiety/ depression) and the visual analogue scale, 5Q-5D-VAS, ranging from 0 to 100.

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Brummer, MD, PhD, Principal Investigator — Örebro University, Sweden
Locations (1):
- Örebro University, Örebro, Sweden